CLINICAL TRIAL: NCT01672619
Title: Nautilus: Dynamic Craniotomy; New Surgical Technique and Preliminary Results
Acronym: Nautilus
Status: Completed | Type: Observational
Sponsor: Nucleo de Plastica Avancada (Network)
Responsible Party: Sponsor
Other Study IDs: npa - 777 - 12
Record Dates: First submitted 2012-08-18; First posted 2012-08-27 (Estimated); Last update posted 2012-08-27 (Estimated); Status verified 2010-06

CONDITIONS: Children With Craniosynostoses
Keywords: craniosynostoses; Osteogenesis Distraction; craniotomy
MeSH Terms: conditions — Craniosynostoses

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- children with craniosynostosis: children with craniosynostosis aged 6 months to 13
  Interventions: Procedure: dynamic craniotomy

INTERVENTIONS:
Procedure: dynamic craniotomy — Surgical technique of craniotomy spiral without detachment of dura mater
  Other Names: craniotomy helicoid; Craniotomy spiral

SUMMARY:
Being the craniostenoses sutural basically a disease, the fact that the brain being trapped in an enclosure that does not have complacency required to accompany their growth constitutes the challenge of treatment, which aims to restore the complacency of the suture and correct the stenotic compensatory cranial deformity.

This paper proposes the combination of a helicoid osteotomy distraction osteogenesis provided by the use of springs distracting.

DETAILED DESCRIPTION:
As demonstrated by some authors, the curved shape of the helix fits perfectly the remodeling of a curved surface as well as the skullcap. If you do not receive fixation, however, trace the helicoid of the bone osteotomy can turn on a spring that can expand or contract depending on the direction of the force that is received. This form of osteotomy was therefore chosen by the authors to induce bone compliance areas of secondary defect that should expand or compress indirectly during the process of dynamic remodeling of primary defect with springs.

ELIGIBILITY:
Inclusion Criteria:

* age between 6 months to 13 years

Exclusion Criteria:

* absence of clinical conditions for the surgical treatment

Ages: 6 Months to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children with craniosynostoses
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2010-06; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Nautilus: dynamic craniotomy; new surgical technique and preliminary results | Up to 3 years
  This study proposes to analyze the cranial remodeling achieved through the use of a dynamic craniotomy, without detachment of the dura mater in cranial deformities caused by craniosynostosis.
cranial remodeling | Up to 3 years
  Quantify the results of cranial remodeling by osteotomy helicoid-shaped Nautilus by clinical and CT in 6 months after the procedure, by 3 surgeons at different times - The skull shape, postoperatively, will be assessed independently by four surgeons, who will use the following scale results: insufficient when there was no attenuation of preoperative deformity, partial, when the correction happened, but was not able to capture all the characteristics of the deformity; appropriate, when there was complete remission of cranial deformity.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Beneficencia Portuguesa de São Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Lauritzen CGK, Davis C, Ivarsson A, Sanger C, Hewitt TD. The evolving role of springs in craniofacial surgery: the first 100 clinical cases. Plast Reconstr Surg. 2008 Feb;121(2):545-554. doi: 10.1097/01.prs.0000297638.76602.de. PMID 18300975